CLINICAL TRIAL: NCT00815308
Title: An Open-labeled Study to Evaluate Efficacy of Combining Erbitux Plus Concurrent Chemo-radiotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Erbitux Combined With Chemo-radiotherapy in Esophageal Squamous Cell Carcinoma
Acronym: EXCEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Hebei Fourth Hospital (Unknown); Jiangsu Cancer Institute & Hospital (Other); RenJi Hospital (Other); The Affiliated Cancer Hospital of Zhengzhou University (Unknown); West China Hospital (Other)
Responsible Party: Jinming Yu, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDRTC-0901
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2009-07

CONDITIONS: Esophageal Cancer
Keywords: Therapeutic; Drug Therapy, combination; Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cetuximab; Paclitaxel; Cisplatin; Radiation; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cetuximab, concurrent chemo-radiotherapy (Experimental): Cetuximab, injection, loading dose400 mg/m^2,(Day1 in Week1) followed by 250 mg/m^2(Day1, every week for Weeks 2-8) Paclitaxel, injection,45 mg/m^2 (Day 1, every week for Weeks 2-8) Cisplatin, injection,20 mg/m^2 (Day 1, every week for Weeks 2-8) radiation therapy, 59.4 Gy, 1.8 Gy/33 fractions,1 fraction daily, Days 1-5 every week for Weeks 2-7, and Days 1-3 for Week 8
  Interventions: Drug: cetuximab (Erbitux); Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: cetuximab (Erbitux) — Cetuximab,injection,loading dose400 mg/m^2,(Day1 in Week1) followed by 250 mg/m^2(Day1, every week for Weeks 2-8)
  Other Names: erbitux
Drug: Paclitaxel — Paclitaxel,injection,loading dose 45 mg/m^2,(Day1 in every week for Weeks 2-8)
Drug: Cisplatin — Cisplatin,injection,loading dose 20 mg/m^2,(Day1 in every week for Weeks 2-8)
Radiation: Radiation — Radiation, External beam therapy, total 59.4 Gy , 33 fractions, 1.8 Gy per fraction.(Day 1-Day 5 in every week 2-week 8).
  Other Names: Conformal Radiotherapy; Intensity Modulated Radiotherapy

SUMMARY:
The purpose of this study is to determine whether the treatment of locally advanced esophageal squamous cell carcinoma (ESCC)with cetuximab in combination with paclitaxel, cisplatin and radiation improve clinical outcomes.

DETAILED DESCRIPTION:
Esophageal cancer is the sixth leading cause of cancer death worldwide.

Over the past 2 decades, well-designed clinical trials have documented the clinical benefits of combination of chemotherapy and radiation for localized esophageal cancer, either as primary therapy or in neoadjuvant setting.

Paclitaxel, a radiation sensitizer, has important single-agent activity in esophageal cancer. Paclitaxel-based chemoradiation has been the framework for the recent Radiation Therapy Oncology Group (RTOG) trials of nonoperative management of esophageal cancer.

Accumulating clinical evidence suggests that epidermal growth factor receptor (EGFR) represents a viable target in the treatment of esophageal cancer. EGFR expression is associated with poor prognosis. Cetuximab, a monoclonal antibody, binds specifically to EGFR on both normal and tumor cells and competitively inhibits the binding of EGF and other ligands, such as transforming growth factor (TGF)-α.

Preclinical models have suggested synergy between cetuximab, paclitaxel, cisplatin and radiation. For patients with locally advanced head and neck cancer, the combination of cetuximab and radiation has demonstrated both response and survival benefit.

With all these, the investigators hypothesize that treatment of locally advanced esophageal squamous cell carcinoma (ESCC)with cetuximab in combination with paclitaxel, cisplatin and radiation may further improve clinical outcomes. This trial results will be important as it may support further studies for setting the new treatment standard for ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients, ≥ 18 years of age
* Histologically confirmed primary (non-recurrent) ESCC fulfilling one of the following criteria (AJCC Staging System)

  * cervical esophageal carcinoma, stage Ⅱ-Ⅲ
  * upper thoracic esophageal carcinoma, stage Ⅱ-Ⅲ, or mid-thoracic esophageal carcinoma, stage Ⅱ-Ⅲ,which is medically unfit for surgery, surgery been refused and patient medically able to tolerate chemo-radiation.
* Evidence of unidimensional measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST).
* ECOG Performance status of 0-1
* Effective contraception for both male and female patients if the risk of conception exists
* Adequate bone marrow reserves: neutrophil (ANC) count ≥ 1500 /mm^3, platelet count ≥ 100,000 /mm^3, hemoglobin ≥ 9 g/dl
* Adequate renal function: serum creatinine ≤ 1.5 mg/dl and/or calculated creatinine clearance ≥ 60 ml/min
* Adequate hepatic function: bilirubin level ≤ 1.5 x ULN, ASAT & ALST ≤ 1.5 x ULN
* Tumor tissue available for KRAS biomarker test
* Signed written informed consent prior to study entry

Exclusion Criteria:

* Previous chest radiotherapy, systemic chemotherapy, and major esophageal surgery
* Concurrent chronic systemic immune therapy, targeted therapy not indicated in this study protocol
* Multiple primary carcinomas of the esophagus
* Pregnancy (confirmed by serum or urine β-HCG) or lactation period;
* Uncontrolled diabetes, hypertension, and severe cardiac or pulmonary disease
* Unable to comprehend the study requirements or who are not likely to comply with the study parameters;
* Distant metastasis
* Second malignancy, except for curable non-melanoma skin cancer, cervical cancer in situ, or malignant disease, free for ≥ 5 years
* Known grade 3 or 4 allergic reaction to any of the study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ming Yu, PH.D, M.D, Study Chair — Shandong Cancer Hospital and Institute
Locations (1):
- Department of Radiation Oncology, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

REFERENCES:
- [Result] Urba SG, Orringer MB, Turrisi A, Iannettoni M, Forastiere A, Strawderman M. Randomized trial of preoperative chemoradiation versus surgery alone in patients with locoregional esophageal carcinoma. J Clin Oncol. 2001 Jan 15;19(2):305-13. doi: 10.1200/JCO.2001.19.2.305. PMID 11208820
- [Result] Kelsen DP, Ginsberg R, Pajak TF, Sheahan DG, Gunderson L, Mortimer J, Estes N, Haller DG, Ajani J, Kocha W, Minsky BD, Roth JA. Chemotherapy followed by surgery compared with surgery alone for localized esophageal cancer. N Engl J Med. 1998 Dec 31;339(27):1979-84. doi: 10.1056/NEJM199812313392704. PMID 9869669
- [Result] Bosset JF, Gignoux M, Triboulet JP, Tiret E, Mantion G, Elias D, Lozach P, Ollier JC, Pavy JJ, Mercier M, Sahmoud T. Chemoradiotherapy followed by surgery compared with surgery alone in squamous-cell cancer of the esophagus. N Engl J Med. 1997 Jul 17;337(3):161-7. doi: 10.1056/NEJM199707173370304. PMID 9219702
- [Result] Walsh TN, Noonan N, Hollywood D, Kelly A, Keeling N, Hennessy TP. A comparison of multimodal therapy and surgery for esophageal adenocarcinoma. N Engl J Med. 1996 Aug 15;335(7):462-7. doi: 10.1056/NEJM199608153350702. PMID 8672151
- [Result] Herskovic A, Martz K, al-Sarraf M, Leichman L, Brindle J, Vaitkevicius V, Cooper J, Byhardt R, Davis L, Emami B. Combined chemotherapy and radiotherapy compared with radiotherapy alone in patients with cancer of the esophagus. N Engl J Med. 1992 Jun 11;326(24):1593-8. doi: 10.1056/NEJM199206113262403. PMID 1584260
- [Result] Raben D, Helfrich B, Bunn PA Jr. Targeted therapies for non-small-cell lung cancer: biology, rationale, and preclinical results from a radiation oncology perspective. Int J Radiat Oncol Biol Phys. 2004;59(2 Suppl):27-38. doi: 10.1016/j.ijrobp.2004.01.054. PMID 15142632
- [Result] Langer CJ. Emerging role of epidermal growth factor receptor inhibition in therapy for advanced malignancy: focus on NSCLC. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):991-1002. doi: 10.1016/j.ijrobp.2003.09.099. PMID 14967461
- [Result] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab, Concurrent Chemo-radiotherapy
Started | 55
Completed | 45
Not Completed | 10
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 0
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab, Concurrent Chemo-radiotherapy
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 57.68 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 45
Region of Enrollment [Number; unit: participants]
  China | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response Rate (RR)
Description: The overall response rate was defined as the numbers of patients with a complete response (CR) or partial response (PR). CR was defined as no target lesion at follow-up computed tomography scan and barium swallow examination 3-6 weeks after completion of chemo-radiation. PR was defined at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 1 to 3 month after therapy
Measure: Number; unit: participants
Arm/Group | Cetuximab, Concurrent Chemo-radiotherapy
Number analyzed (Participants) | 55
participants | 44

2. Secondary Outcome: Number of Participants With Toxicity
Description: All patients were regularly monitored for possible adverse events, which were graded according to National Cancer Institute Common Toxicity Criteria version 3.0.
Time Frame: Every week during treatment and 1 month after therapy
Measure: Number; unit: participants
Arm/Group | Cetuximab, Concurrent Chemo-radiotherapy
Number analyzed (Participants) | 55
participants | 55

3. Secondary Outcome: Participants With Overall Survival (OS) at 1 Year
Time Frame: 1 year from the date of diagnosis
Reporting Status: Not Posted, anticipated posting 2011-08
Measure: Number; unit: participants

4. Secondary Outcome: Participants With Overall Survival (OS) at 3 Year
Time Frame: 3 year from the date of diagnosis
Reporting Status: Not Posted, anticipated posting 2013-08
Measure: Number; unit: participants

5. Secondary Outcome: Participants With Progression Free Survival (PFS)
Time Frame: Recurrence or metastasis from the date of diagnosis
Reporting Status: Not Posted, anticipated posting 2013-08
Measure: Number; unit: participants

6. Secondary Outcome: Number of Participants With K-ras Gene Mutation
Description: DNA was extracted from tumor specimens.Screened for the presence of KRAS codon 12 and 13 mutations using a PCR clamping and melting curve technique. PCR amplification of the wild-type KRAS sequence was suppressed in this process by the incorporation in the reaction mix of a locked nucleic-acid oligomer16 spanning codons 12 and 13 of the KRAS gene. Post-PCR hybridization and melting curve analysis using fluorescently tagged oligonucleotides incorporated in the original PCR reaction permitted the identification and discrimination of distinct KRAS codon 12 and 13 missense mutations.
Time Frame: 07/29/2010-09/30/2010
Measure: Number; unit: participants
Arm/Group | Cetuximab, Concurrent Chemo-radiotherapy
Number analyzed (Participants) | 55
participants | 53

ADVERSE EVENTS:
Arm/Group | Cetuximab, Concurrent Chemo-radiotherapy
Serious Adverse Events (participants affected / at risk) | 2/55
Other Adverse Events (participants affected / at risk) | 38/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab, Concurrent Chemo-radiotherapy (N=55)
esophago-tracheal fistula (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.81% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab, Concurrent Chemo-radiotherapy (N=55)
Hepatic Functional Lesion (Hepatobiliary disorders) | 2 (2)
Granulocytopenia (Blood and lymphatic system disorders) | 18 (18)
Skin Eruption (Skin and subcutaneous tissue disorders) | 1 (1)
granlopenia (Blood and lymphatic system disorders) | 4 (4)
radiodematitis (Skin and subcutaneous tissue disorders) | 4 (4)
mucositis (Skin and subcutaneous tissue disorders) | 7 (7)
radioacitvity esophagitis (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No